CLINICAL TRIAL: NCT01534351
Title: A Phase III, Randomized Clinical Trial to Study the Safety and Efficacy of MK-906 (Finasteride) and Tamsulosin Administered Either Alone or Concomitantly in Patients With Benign Prostatic Hyperplasia (BPH)
Brief Title: Comparison of Finasteride and Tamsulosin for Treatment of Benign Prostatic Hyperplasia (BPH) (MK-0906A-149 AM2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0906A-149
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Finasteride; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Finasteride (Experimental): Finasteride 5 mg taken orally once daily and tamsulosin-matching placebo taken orally once daily for 12 months. The tamsulosin-matching placebo will be taken approximately one half hour following the same meal each day. Medications may be taken separately or together.
  Interventions: Drug: Finasteride; Drug: Tamsulosin-matching placebo
- Tamsulosin (Active Comparator): Tamsulosin 0.2 mg taken orally once daily and finasteride-matching placebo taken orally once daily for 12 months. The tamsulosin will be taken approximately one half hour following the same meal each day. Medications may be taken separately or together.
  Interventions: Drug: Tamsulosin; Drug: Finasteride-matching placebo
- Finasteride and Tamsulosin (Experimental): Finasteride 5 mg orally once daily and tamsulosin 0.2 mg orally once daily for 12 months, taken concomitantly. The tamsulosin will be taken approximately one half hour following the same meal each day. Medications may be taken separately or together.
  Interventions: Drug: Finasteride; Drug: Tamsulosin

INTERVENTIONS:
Drug: Finasteride — Finasteride 5 mg oral tablet taken once daily.
  Other Names: Proscar®
  Arms: Finasteride; Finasteride and Tamsulosin
Drug: Tamsulosin — Tamsulosin 0.2 mg oral capsule taken once daily.
  Other Names: Flomax®
  Arms: Finasteride and Tamsulosin; Tamsulosin
Drug: Finasteride-matching placebo — Matching placebo to finasteride 5 mg oral tablet taken once daily.
  Arms: Tamsulosin
Drug: Tamsulosin-matching placebo — Matching placebo to tamsulosin 0.2 mg oral capsule taken once daily.
  Arms: Finasteride

SUMMARY:
This study is designed to compare safety and efficacy of monotherapy finasteride to combination therapy (finasteride and tamsulosin) in Asian men with benign prostatic hyperplasia (BPH) who are at least 50 years of age or older. The primary hypotheses are that concomitantly-dosed finasteride 5 mg and tamsulosin 0.2 mg will be superior with respect to BPH symptoms compared to monotherapy with finasteride 5 mg as measured by change from baseline on the International Prostate Symptoms Score (IPSS) and will be superior with respect to prostate volume reduction compared to montherapy with tamsulosin 0.2 mg as measured by percent change from baseline in prostate volume.

ELIGIBILITY:
Inclusion Criteria:

* Possess a clinical diagnosis of BPH.
* Able to read, understand, and complete the study questionnaire.

Exclusion Criteria:

* History or recurrent evidence of any condition, therapy, lab abnormality or other circumstance that might confound the results of the study, or interfere with participation for the full duration of the study.
* History of malignancy ≤ 5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer, including prostate cancer of any duration, evidence or suspicion of prostate cancer on a previous biopsy.
* History of prostatic surgery or other invasive procedures to treat BPH or history of bladder neck obstruction, bladder cancer, and/or pelvic irradiation, urinary incontinence, recurrent urinary tract infection, urethral stricture, or bacterial prostatitis.
* History of acute urinary retention (ie, inability to fully empty bladder).
* Had invasive urinary bladder procedures (ie, cystoscopy) within 7 days prior to screening.
* Had phytotherapy within 2 weeks of screening and may need phytotherapy during the study.
* History of low blood pressure (orthostatic hypotension, hypotension [supine blood pressure less than 90/70 mm Hg]), unstable angina, or a cardiovascular or cerebral vascular event (ie, transient ischemic attack [TIA], stroke) within the previous 3 months prior to enrollment, OR a history of dizziness, vertigo or any other typical signs and symptoms of low blood pressure.
* Recent history (ie, within the past year) or active addiction, abuse, misuse of and/or dependence on drugs and/or alcohol.
* Use of herbal therapies that may impact the study (eg, Saw Palmetto) within 2 weeks of screening and/or is predicted to need herbal therapies during the study. Individuals currently taking herbal therapies may be eligible for study if willing to complete a 2-week washout period.
* Use of finasteride or a drug with a similar action during the 12 months prior to study screening. Individuals treated for short periods with 5-alpha reductase inhibitors (5ARIs) or drugs with antiandrogenic properties within 12 months of screening may be eligible for study.
* Use of a non-approved (investigational) drug within the last 4 weeks prior to enrollment, or current participation in another clinical study.
* Allergic or intolerant to finasteride and/or tamsulosin.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2013-11-18 (Actual); Study Completion 2013-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0906A-149&kw=0906A-149&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to early study discontinuation, 3 sites were initiated and screened a total of 8 participants. Of the 8 participants, one participant was randomized to finasteride 5 mg once daily for 39 days.
Groups:
- Finasteride: Finasteride 5 mg taken orally once daily and tamsulosin-matching placebo 0.2 mg taken orally once daily for 12 months. The tamsulosin-matching placebo will be taken approximately one half hour following the same meal each day. Medications may be taken separately or together.
- Tamsulosin: Tamsulosin 0.2 mg taken orally once daily and finasteride-matching placebo 5 mg taken orally once daily for 12 months. The tamsulosin will be taken approximately one half hour following the same meal each day. Medications may be taken separately or together.
Period: Overall Study
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Study Terminated Early | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 1 |  |  | 1
  >=65 years | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  | 0
  Male | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS)
Description: The IPSS is a self-administered questionnaire used to measure the severity of lower urinary tract symptoms among men suspected of having symptomatic Benign Prostatic Hyperplasia (BPH). The IPSS consists of 8 questions (7 urinary symptom questions + 1 quality of life question). The 7 symptom questions inquire about frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying and urgency. Each of the 7 questions has an ordered categorical response frame scored from 0 (not at all) to 5 (almost all the time). The total score is the sum of the 7 items and therefore has a range of 0 to 35. Higher scores indicate higher symptom severity. The quality of life question is a single global question rated on a scale of 0 (delighted) to 6 (terrible) asking the participant to rate how they feel about their current urinary symptom status. The IPSS-QoL question is not used in the calculation of the total symptom score.
Time Frame: Baseline and Month 12
Population: Full Analysis Set (FAS) - population consists of all randomized participants who received at least one dose of study treatment, at least one post-randomization observation for the analysis endpoint, and baseline data for those analyses that require baseline data. As only one participant was randomized in the study, no analyses were performed.
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Percent Change From Baseline in Prostate Volume
Description: Prostate volume was assessed by trans-rectal ultrasound (TRUS).
Time Frame: Baseline and Month 12
Population: as for outcome 1
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product.
Time Frame: Up to 54 weeks
Measure: Number; unit: Participants
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin
Number analyzed (Participants) | 1 | 0 | 0
Participants | 0 |  |

4. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event
Description: as for outcome 3
Time Frame: Up to 52 weeks
Population: All Participants as Treated (APaT) - population consists of all randomized participants who received at least one dose of study treatment. As only one participant was randomized in the study, no analyses were performed.
Measure: Number; unit: Participants
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin
Number analyzed (Participants) | 1 | 0 | 0
Participants | 0 |  |

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Arm/Group | Finasteride | Tamsulosin | Finasteride and Tamsulosin
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The trial was terminated for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.